CLINICAL TRIAL: NCT05718583
Title: A Pilot Proof of Concept Study of the Effects of Administration of a Short Chain Fatty Acid (SCFA) Supplement in Rheumatoid Arthritis Inadequate Responders (EASi-RAIR)
Brief Title: Effects of Administration of SCFA in Rheumatoid Arthritis Inadequate Responders
Acronym: EASi-RAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-01526
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Short Chain Fatty Acid; Butyrate; Microbiome; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Butyrates; Butyric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RA Patients who are Inadequate Responders to Current RA Treatment (Experimental): Oral butyrate will be taken at 1000 mg three times daily with meals by RA patients who have active disease and are currently taking methotrexate (MTX) at prescriber's recommended dose. There will be no dose escalation of the study supplement. Clinical data to assess for adverse events, stool, urine samples and peripheral blood will be collected at baseline, 1 month, and with an optional 2-month time-point.
  Interventions: Dietary Supplement: Butyrate

INTERVENTIONS:
Dietary Supplement: Butyrate — Participants will self-administer the oral Short Chain Fatty Acid (SCFA) Butyrate supplement three times daily with meals for up to 2 months. The minimum duration necessary for an "evaluable" participant will be 2 weeks of SCFA supplementation.
  Other Names: Butyrate; butyric acid

SUMMARY:
This study is a pilot, proof of concept study to determine the effects of administering an oral short-chain fatty acid (SCFA) supplement to Rheumatoid Arthritis (RA) patients with inadequate response to methotrexate (MTX). The study will include up to 35 participants to obtain a sample size of at least 25 participants taking the oral supplement. The researchers hypothesize that oral SCFA will change the participants' gut microbiome and regulatory immune responses. Clinical data to assess for adverse events, stool, urine samples and peripheral blood will be collected at baseline, 1 month, and with an optional 2 month time-point. Fecal microbiome will be analyzed. Adaptive immune responses will be analyzed from participant blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of RA meeting 2010 ACR/EULAR for RA and/or treating MD diagnosis
2. Inadequate response to MTX per treating MD at maximum tolerated dose.
3. Able and willing to provide written informed consent prior to any study specific procedures
4. Age 18 years and above at time of enrollment
5. Subjects not excluded based on race or ethnicity

Exclusion Criteria:

1. Participants who are pregnant or are currently breastfeeding
2. History of sensitivity to study compound or any of their excipients
3. Previous intolerance to SCFA or related compounds
4. Current antibiotic treatment (within 3 months of screening) at discretion of PI
5. Current consumption of probiotics (within 3 months of screening) at discretion of PI
6. Severe hepatic impairment (eg, ascites and/or clinical signs of coagulopathy)
7. Renal failure (eGFR <30 or requiring dialysis) by history
8. History of other autoimmune disease at discretion of PI
9. Current immunodeficiency state (e.g., cancer, HIV, others)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Microbiome Alpha Diversity | Baseline, Month 1 Post-Treatment Initiation
  Measured by Shannon diversity index.

SECONDARY OUTCOMES:
Change in Serum SCFA Concentration | Baseline, Month 1 Post-Treatment Initiation
  Measured via participant blood draws.
Change in Fecal SCFA Concentration | Baseline, Month 1 Post-Treatment Initiation
  Measured via participant stool samples.
Change in Peripheral Regulatory T Cell Concentration | Up to Month 1 Post-Treatment Initiation
  Measured via participant blood draws.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Blank, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health Orthopedic Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [Rebecca.blank@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Rebecca.blank@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.